CLINICAL TRIAL: NCT00436358
Title: Implementation of Hospital-based Active Surveillance Procedures for Vaccine Safety Monitoring at IMSS Hospitals With Pediatric Medical Care in Mexico
Brief Title: Implementing Hospital-based Active Surveillance Procedures for Vaccine Safety Monitoring at IMSS Hospitals in Mexico
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Other Study IDs: 106175
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Intussusception; LRTI-related Post Neonatal Deaths
Keywords: Mexico; Intussusception; Epidemiology
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (5):
- Group A: IS case deemed children
  Interventions: Other: Not applicable: none
- Group B: LRTI-related post-neonatal deaths deemed Children
  Interventions: Other: Not applicable: none
- Group C: A random sample of children from an annual birth cohort within the electronic IMSS dataset
  Interventions: Other: Not applicable: none
- Group D: All children from a single annual birth cohort with IS identified in their electronic IMSS data
  Interventions: Other: Not applicable: none
- Group E: A sample of children from the electronic IMSS dataset selected to match the selected IS cases on age, gender, and hospital of birth.
  Interventions: Other: Not applicable: none

INTERVENTIONS:
Other: Not applicable: none — Please refer to the detailed description section

SUMMARY:
This is an epidemiology study designed to implement hospital-based active surveillance for intussusception (IS) in children <1 year of age and lower respiratory tract infection (LRTI)-related deaths among children between 29 days and 1 year of age in Mexico. An existing linked database of the "Instituto Mexicano del Seguro Social (IMSS)" will be used. The study described in this protocol is a pilot study, which will evaluate the methodology to be used in a later Post-Marketing Surveillance (PMS) study.

The planned epidemiology study will be conducted in IMSS hospitals and potentially use the IMSS database to re-capture potential cases of IS and fatal cases and as a source of matched case controls. The purpose of this project is to complement this data link system with an active surveillance system for IS - in order to assess the feasibility of using the IMSS data system by generating results that provide scientific validity. Such comprehensive (passive and active) surveillance systems will facilitate the post licensure safety profile evaluation of vaccines such as a vaccine against rotavirus diarrhoea.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The main aim of this pilot study is to allow for the implementation of active hospital-based surveillance for IS in children <1 year of age in IMSS hospitals with pediatric medical care, and LRTI-related post-neonatal deaths among children between 29 days and 1 year of age participating in the IMSS system. Surveillance will be conducted in each of the approximately 230 IMSS hospitals with pediatric medical care (tertiary care and secondary care hospitals), which have 40 million affiliates and an annual birth cohort of 575,000.

During the pilot phase the completeness and validity of electronic vaccination and demographic data contained in the IMSS dataset will be assessed to determine whether or not these data will be used during the actual post licensure study implementation. Study participation for database validation will include parental/guardian/legal representative interview and review of vaccination records.

Study staff at each of the approximately 230 IMSS hospitals will review medical records daily for potential cases of IS in children <1 year of age.

Medical records of potential IS cases will be reviewed to determine eligibility, in terms of IS, based on the Brighton criteria Parents/guardians/legal representative of definite IS cases will be contacted by study staff to recruit their child into the study.

After the informed consent is signed, the parental/guardian interview will be conducted.

Additional medical information will be collected through medical record review during hospitalization and after the child has been discharged.

A central Information Coordinator (IMSS staff member) will perform monthly reviews of the IMSS database to search for definite IS cases.

A cross-check will be performed with IMSS database to identify definite IS cases not yet enrolled. In that situation, parents/guardians/legal representative will be contacted by study staff to recruit their child into the study. Either in-hospital interviews or in-home interviews will be arranged to collect data.

Study staff will perform the same review as above but for LTRI-related deaths in children between 29 days and 1 year of age. They will also review morgue records for LRTI-related deaths.

A central Information Coordinator (IMSS staff member) will perform monthly reviews of the IMSS database for post-neonatal LRTI-related deaths.

Study staff will contact the parents/guardians/legal representative of the deceased child to explain the study and request enrollment.

After informed consent is obtained, an interview will be conducted with parents/guardians/legal representative.

IMSS medical records will be reviewed by study staff. All LTRI related post-neonatal deaths will be reported to the Principal Investigator (PI) and to the Safety Review Expert Committee (SReC).

The SReC, which is completely independent from GSK Biologicals, will assign causes of death (CoD) for all enrolled LTRI-related post-neonatal death cases.

All definite IS cases and LTRI related post-neonatal fatalities will be reported to the GSK local operating company within 24 hours of identification. In addition all SAEs, deemed to be related to a GSK vaccine will be reported based on discharged diagnosis only.

The completeness of key demographic data (date of birth, hospital of birth, gender, and residential address) will be assessed for a sample of children in the IMSS dataset in a single annual birth cohort.

A random sample (N=1,200) of children from a single annual birth cohort will be selected from the IMSS dataset for verification of demographic data and vaccination history (the selection process will continue until informed consent has been obtained for a total of 1,200 children). In-home interviews will be conducted with parents/guardians/legal representative of all 1200 subjects to gather demographic and vaccination history (EPI card - Cartilla Nacional de Vacunacion).

Demographic data collected in the interview will be compared to that in the IMSS dataset.

Vaccine history (two doses of DTP) collected from the EPI vaccination cards will be compared to that in the IMSS dataset. The agreement for DTP will be assessed.

All IS episodes in a single annual birth cohort of children in the IMSS dataset will be identified. Data necessary for selection of matched controls (date of birth, hospital of birth, and gender) will be extracted for these children.

Five controls for identified IS cases will be selected from the IMSS dataset based on the ability to fulfil the matching criteria. Statistics on the number of matched controls and the quality of the match will be assessed by IMSS and Rixensart statisticians.

Primary outcome measure: occurrence of IS by passive (IMSS database) and active (RDE) surveillance and of LRTI-related post-neonatal deaths by passive and active surveillance.

Secondary outcome measure: demography data of IMSS affiliate, from IMSS record and parent interview; DTP history from IMSS dataset and EPI

ELIGIBILITY:
Inclusion Criteria:

An IS case deemed eligible for the study must meet the following criteria:

* Subject is an IMSS affiliate
* Subject is being treated/has been treated at one of the IMSS hospitals/medical facilities with IS during the study period.
* Male or female child is <1 year of age at the time of diagnosis of the IS
* Subject is diagnosed with definite IS
* Written informed consent for definite IS cases is obtained from the parent/guardian/legal representative of the subject.
* Only subjects who the investigator believes will meet the requirements of the protocol should be enrolled in the study.

A death deemed eligible for the study must meet the following criteria:

* Subject is an IMSS affiliate
* Death certificate is available
* Male or female child between 29 days and 1 year of age, at the time of death
* Post-neonatal LRTI-related death occurred during the study period
* Written informed consent is obtained from the parent/guardian/legal representative of the subject.

For a child to be included in the random sample selected from the IMSS dataset must meet the following criteria:

* Subject is an IMSS affiliate.
* Male or female child belonging to the annual birth cohort selected for the evaluation.
* Written informed consent is obtained from the parent/guardian/legal representative of the subject.
* Subject did not die.
* Subject currently lives in Mexico.

IS Cases Selected from IMSS Dataset must meet the following criteria:

* Subject with an IS identified in the IMSS dataset.
* Male or female child is <1 year of age at the time of diagnosis of the IS (patient becomes ineligible on the day of their first birthday).
* Subject belongs to the annual birth cohort selected for the evaluation.

Children Selected as Controls for Matched Assessment

• subject matched to a case by gender, hospital of birth and date of birth as described above.

Exclusion Criteria:

For a child to be included as a matched control:

* subject is dead
* subject is not currently living in Mexico
* subject experienced an IS episode recorded in the IMSS database.

Exclusion criteria for enrollment: none

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: IMSS hospitals with pediatric medical care in Mexico
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of IS by passive (IMSS database) and active (RDE) surveillance | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.
Occurrence of LRTI-related post-neonatal deaths by passive surveillance (IMSS database) and active surveillance (RDE) | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.
Key demographic data (date of birth, hospital of birth, gender, and residential address) of IMSS affiliate | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.
Demographic data (date of birth, hospital of birth, gender, and residential address) from the electronic IMSS record of IMSS affiliate | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.
Demographic data (date of birth, hospital of birth, gender, and residential address) collected from parent/guardian/legal representative/guardian interview | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.
Vaccination history (DTP) from electronic IMSS dataset of IMSS affiliate | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.
Vaccination history (DTP) from EPI cards of IMSS affiliate. | Approx 3 months to initiate the active surveillance systems in approx 230 hospitals. Three additional months, after implementation, may be required to generate some baseline data as well as to start generating database validation results.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mexico City, Mexico